CLINICAL TRIAL: NCT00089960
Title: An Open Label Study of AMG 706 in Subjects With Advanced Gastrointestinal Stromal Tumors (GISTs) Who Developed Progressive Disease or Relapsed While on Imatinib Mesylate
Brief Title: Study of AMG 706 in Subjects With Advanced Gastrointestinal Stromal Tumors (GISTs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040110
Expanded Access: Available
Record Dates: First submitted 2004-08-18; First posted 2004-08-20 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Gastrointestinal Cancer
Keywords: GIST
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — motesanib diphosphate

ARMS (1):
- Arm (Other): AMG 125 mg daily continuously
  Interventions: Drug: AMG 706

INTERVENTIONS:
Drug: AMG 706 — AMG 706 125 mg daily for 48 weeks, or until progressive disease or unacceptable toxicity.

SUMMARY:
This study will determine the safety and effectiveness of AMG 706 in patients with advanced GIST.

DETAILED DESCRIPTION:
Expanded Access: Amgen provides expanded access for this clinical trial. Contact the Amgen Call Center (866-572-6436) for more information.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years;
* Disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) during previous treatment with imatinib mesylate at least 600 mg daily for at least 8 weeks, as per two independently assessed prestudy computerized tomography (CT) scans;
* Presence of at least one measurable (per RECIST)
* Progressing tumor lesion not previously treated with radiotherapy or embolization and evaluable by CT scan or magnetic resonance imaging (MRI);
* Karnofsky performance status ≥ 60;
* imatinib treatment terminated at least 7 days before study day 1;
* Adequate hepatic, renal, and cardiac function.

Exclusion criteria:

* Prior malignancy (other than GIST, in situ cervical cancer, or basal cell cancer of the skin) unless treated with curative intent and without evidence of disease for ≥ 3 years; cardiac disease including myocardial infarction, unstable angina, and congestive heart failure (New York Heart Association class > II),
* uncontrolled hypertension (systolic > 145 mmHg or diastolic > 85 mmHg),
* History of arterial thrombosis or deep vein thrombosis (including pulmonary embolus) within 1 year of study day 1;
* Absolute neutrophil count < 1.5x109/L, platelet count < 100x109/L, hemoglobin < 9.0 g/dL;
* Prior treatment with motesanib diphosphate or other KIT (except imatinib) or VEGF inhibitors.
* The study was approved by the institutional review board of each participating institution, and all patients provided written informed consent before any study-related procedures were performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2004-10; Primary Completion 2006-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate as defined using modified RECIST criteria. | 48 weeks treatment or until progressive disease, or unacceptable toxicity

SECONDARY OUTCOMES:
Progression-free survival | time from randomization to progressive disease
Overall survival | time to death
Time to progression | time from response to progressive disease
Time to response | time from first treatment to response
Patient-reported outcomes | quality of life
Use of opioid analgesics after minimal 6 months treatment | narcotics usage during study
Objective response by PET and tumor size/density changes at week 8 | response rate at week 8
Objective response by size changes and/or target tumor density changes at week 8 | response rate at week 8
Safety Endpoints: Incidence of adverse events (including all, serious, grade 3, grade 4 and treatment related) | for duration of study
Duration of response | time to respone to progression
Palliative response | amelioration of symptoms
Pharmacokinetic Endpoints: 1. The AMG 706 PK parameters (Cmax, t1/2, AUC0-24, C24); 2. To explore the PK/PD relationships | during specific study timepoints

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Benjamin RS, Schoffski P, Hartmann JT, Van Oosterom A, Bui BN, Duyster J, Schuetze S, Blay JY, Reichardt P, Rosen LS, Skubitz K, McCoy S, Sun YN, Stepan DE, Baker L. Efficacy and safety of motesanib, an oral inhibitor of VEGF, PDGF, and Kit receptors, in patients with imatinib-resistant gastrointestinal stromal tumors. Cancer Chemother Pharmacol. 2011 Jul;68(1):69-77. doi: 10.1007/s00280-010-1431-9. Epub 2010 Sep 14. PMID 20838998
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_63_AMG_706_20040110.pdf